CLINICAL TRIAL: NCT01881035
Title: Treatment of Resistant Hypertension by Renal Sympathetic Denervation in Patients Undergoing Dialysis Therapy
Acronym: TreatDialRDN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting of the whole study population not possible.
Sponsor: Turku University Hospital (Other Government)
Collaborators: Oulu University Hospital (Other); Satakunta Central Hospital (Other); Central Finland Hospital District (Other); Vaasa Central Hospital, Vaasa, Finland (Other)
Responsible Party: Principal Investigator, Juhani Koistinen, Professor in Medicine Turku University, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCH Heart Station 10; TreatDialRDN (II) (Other: Turku University Finland)
Record Dates: First submitted 2013-06-14; First posted 2013-06-19 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Hypertension Secondary to Renal Disease
Keywords: Hypertension; End stage renal disease
MeSH Terms: conditions — Hypertensive Nephropathy; Hypertension; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Renal nerve denervation (Experimental): Renal nerve denervation
  Interventions: Procedure: Renal nerve denervation

INTERVENTIONS:
Procedure: Renal nerve denervation — Renal nerve denervation is performed by catheter ablation of renal arteries influencing the sympathetic nerves.

SUMMARY:
The study is designed to investigate the efficacy of renal nerve denervation in treating drug-resistant hypertension in patients with end stage renal disease.

DETAILED DESCRIPTION:
Drug resistant hypertension is very common in end stage renal disease treated by dialysis. The prevalence of hypertension has been evaluated to be over 50% and up 80%. In this patient group mortality figures are high because of cardiovascular diseases which are complications of hypertension. Renal nerve denervation is a new intervention to treat hypertension. By applying radiofrequency pulses to the renal arteries, the nerves in the vascular wall (adventitia layer) can be denervated. This causes reduction of renal sympathetic afferent and efferent activity and blood pressure can be decreased. The technique and its efficacy in end stage renal disease has not been systematically studied. There are case reports which have showed promising responses to denervation. In the present study 30 patients over 18 years are planned undergo renal denervation if the medical treatment (three different drugs including diuretics) has failed to decrease blood pressure sufficiently(160/100mmHg). The failure of medical treatment will be documented by ambulatory blood pressure measurements. After renal nerve denervation a two year follow-up of patients with ambulatory blood pressure measurements will be organized. The blood pressures before and after denervation are compared and the quality of life of the patients is evaluated by questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* patients with end stage renal disease and drug-resistant blood pressure.

Exclusion Criteria:

* pregnancy
* secondary hypertension
* unstable coronary artery disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of blood pressures before and after intervention | 2 years

SECONDARY OUTCOMES:
Quality of life | 2 years

OTHER OUTCOMES:
12-lead ECG changes | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Vaasa Central Hospital, Vaasa, Finland

REFERENCES:
- [Derived] Pietila-Effati PM, Salmela AK, Niemi RT, Ylitalo AS, Koistinen MJ. Renal sympathetic denervation in treating drug-resistant hypertension in a patient on hemodialysis. J Hypertens. 2016 Feb;34(2):368-70. doi: 10.1097/HJH.0000000000000802. PMID 26867061